CLINICAL TRIAL: NCT05407402
Title: Examination of the Effect of Laughter Yoga on Pain and Comfort in Individuals Diagnosed With Migraine
Brief Title: Laughter Yoga on Pain and Comfort in Individuals Diagnosed With Migraine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Osmaniye Korkut Ata University (Other)
Responsible Party: Principal Investigator, Kevser Sevgi Ünal Aslan, assistant professor, Osmaniye Korkut Ata University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Korkut Ata Unıversity
Record Dates: First submitted 2022-05-20; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Pain, Head
Keywords: laughter yoga,; funny videos,; migraine,; pain,; comfort
MeSH Terms: conditions — Headache; Migraine Disorders; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- laughter yoga (Experimental): laughter yoga
  Interventions: Behavioral: laughter yoga practice
- funny videos, (Experimental): funny videos,
  Interventions: Behavioral: watching funny videos
- control (No Intervention): control group. routine nursing care will be applied.

INTERVENTIONS:
Behavioral: laughter yoga practice — To reduce the pain and increase the comfort of individuals diagnosed with migraine with these planned interventions.
  Arms: laughter yoga
Behavioral: watching funny videos — To reduce the pain and increase the comfort of individuals diagnosed with migraine with these planned interventions.
  Arms: funny videos,

SUMMARY:
In individuals diagnosed with migraine, laughter yoga will be performed for 45 minutes, 3 times a week for 1 month. the other application group will watch funny videos for 45 minutes, 3 times a week for 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Being older than 18 years of age
* Having been diagnosed with migraine for at least one year
* Having no mental disability

Exclusion Criteria:

* individuals using pain relievers
* individuals who have done laughter yoga before

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-15 (Estimated)

PRIMARY OUTCOMES:
Laughter yoga changes pain | 2 month
  Visual Pain Scale:
  The pain scores of the patients will be measured after the pre-test and the 4th week using the visual pain scale.
Laughter yoga changes comfort. | 2 month
  The General Comfort Scale The General Comfort Scale scores of the patients will be measured after the pre-test and the 4th week using the comfort scale.

OTHER OUTCOMES:
Watching funny videos changes pain | 2 month
  Visual Pain Scale:
  The pain scores of the patients will be measured after the pre-test and the 4th week using the visual pain scale.
Watching funny videos changes comfort. | 2 month
  The General Comfort Scale The General Comfort Scale scores of the patients will be measured after the pre-test and the 4th week using the comfort scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Aksaray University, Aksaray, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
may be published at the discretion of the authors, provided appropriate justifications are provided.